CLINICAL TRIAL: NCT00395070
Title: A Phase 3 Clinical Trial to Evaluate the Safety and Efficacy of Treatment With 2 mg Intralesional Allovectin-7® Compared to Dacarbazine (DTIC) or Temozolomide (TMZ) in Subjects With Recurrent Metastatic Melanoma
Brief Title: A Phase 3 Pivotal Trial Comparing Allovectin-7® Alone vs Chemotherapy Alone in Patients With Stage 3 or Stage 4 Melanoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LX01-315
Record Dates: First submitted 2006-10-31; First posted 2006-11-02 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2013-09

CONDITIONS: Metastatic Melanoma
Keywords: Melanoma; DTIC; TMZ; Stage 3; Stage 4; Metastatic; Metastatic Melanoma (Stage 3, Stage 4 Melanoma)
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis | interventions — Allovectin-7; Dacarbazine; Temozolomide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Arm (Experimental): Allovectin-7® 2 mg intralesional injection into a single lesion weekly for six consecutive weeks, repeated beginning after each 8th week.
  Interventions: Biological: Allovectin-7®
- Control Arm (Active Comparator): DTIC 1000 mg/m2 intravenous infusion over 60 minutes, repeated every 28 days, OR TMZ 150 to 200 mg/m2 orally once daily for five consecutive days, repeated every 28 days.
  Interventions: Drug: Dacarbazine (DTIC); Drug: Temozolomide (TMZ)

INTERVENTIONS:
Biological: Allovectin-7® — Allovectin-7® 2 mg intralesional injection into a single lesion weekly for six consecutive weeks, repeated beginning after each 8th week.
  Arms: Treatment Arm
Drug: Dacarbazine (DTIC) — 1000 mg/m2 intravenous infusion over 60 minutes, repeated every 28 days, OR
  Arms: Control Arm
Drug: Temozolomide (TMZ) — 150 to 200 mg/m2 orally once daily for five consecutive days, repeated every 28 days.
  Arms: Control Arm

SUMMARY:
To compare the safety and efficacy of Allovectin-7® versus Dacarbazine (DTIC)or Temozolomide (TMZ) in subjects with recurrent stage 3 or stage 4 melanoma.

DETAILED DESCRIPTION:
Eligible patients will have a 66% chance of receiving Allovectin-7® alone (an investigational product designed to train your body's immune system to recognize and destroy tumor cells) vs. a 33% chance of receiving standard chemotherapy (either dacarbazine or temozolomide). The treatment course recommended for patients who receive Allovectin-7® is a minimum of 16 weeks. Each cycle will consist of weekly injections of Allovectin-7® alone for six weeks followed by two weeks of observation and assessments. For patients who receive the chemotherapy alone, their treatment course will follow standard dosing. During the trial all patients' tumors will be closely monitored. Patients whose melanoma does not clinically progress will be encouraged to continue on the treatment and be assessed for up to two years.

ELIGIBILITY:
Inclusion Criteria (Potential study participants must meet the following criteria):

* Confirmed Stage 3 or Stage 4 melanoma that may have had previous treatment via surgery, radiation or biologic drugs (typically Interferon Alpha or Interleukin-2)
* At least 1 melanoma tumor that is 1cm x 1cm or greater in size (about the size of a dime) and can be injected
* Normal blood chemistries and blood cell counts
* At least 18 years old and able and willing to provide informed consent to participate

Exclusion Criteria (Potential study participants will not be eligible with the following):

* Previous chemotherapy treatment for melanoma
* Melanoma lesions in the brain or liver (however, lesions in the lungs are allowed)
* If surgical removal of all lesions would be possible and could be curative
* Any melanoma tumors greater than 10cm x 10cm in size
* Known condition resulting in a suppressed immune system
* Female subjects who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2006-10; Primary Completion 2012-03 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
To compare the overall response rate at ≥24 weeks after randomization in the Allovectin-7® arm versus the control (DTIC/TMZ) arm. | After all 375 subjects are enrolled

SECONDARY OUTCOMES:
To investigate the safety/tolerability of Allovectin-7® in comparison to DTIC/TMZ. | After all 375 subjects are enrolled
To investigate the effect of Allovectin-7® in comparison to DTIC-TMZ on overall survival. | After all 375 subjects are enrolled

CONTACTS AND LOCATIONS:
Overall Officials: Linda Strause, PhD, Study Director — Vical
Locations (88):
- United States (27):
  - Location #40, Tucson, Arizona
  - Location #9, Little Rock, Arkansas
  - Location #1, Bakersfield, California
  - Location #24, San Diego, California
  - Location #36, San Diego, California
  - Location #47, San Francisco, California
  - Location #16, Denver, Colorado
  - Location #11, Lakeland, Florida
  - Location #7, Chicago, Illinois
  - Location #33, Chicago, Illinois
  - Location #20, Louisville, Kentucky
  - Location #35, Baltimore, Maryland
  - Location #4, Kansas City, Missouri
  - Location #19, St Louis, Missouri
  - Location #38, Hackensack, New Jersey
  - Location #8, Montclair, New Jersey
  - Location #87, Albuquerque, New Mexico
  - Location #41, Cincinnati, Ohio
  - Location #23, Cleveland, Ohio
  - Location #34, Portland, Oregon
  - Location #12, Bethlehem, Pennsylvania
  - Location #97, Providence, Rhode Island
  - Location #28, Dallas, Texas
  - Location #117, Houston, Texas
  - Location #27, Salt Lake City, Utah
  - Location #26, Salt Lake City, Utah
  - Location #32, Seattle, Washington
- Belgium (2):
  - Location #55, Brussels
  - Location #63, Liège
- Brazil (8):
  - Location #102, Itaquera, São Paulo
  - Location #99, Belo Horizonte
  - Location #101, Curitiba
  - Location #104, Ijuí
  - Location #100, Lajeado
  - Location #103, Porto Alegre
  - Location #105, Rio de Janeiro
  - Location #106, São Paulo
- Canada (3):
  - Location #37, Calgary, Alberta
  - Location #88, Winnipeg, Manitoba
  - Location # 75, Ottawa, Ontario
- France (9):
  - Location #110, Bordeaux
  - Location #112, Lyon
  - Location #113, Marseille
  - Location #114, Montpellier
  - Location #109, Nantes
  - Location #66, Paris
  - Location #74, Paris
  - Location #115, Toulouse
  - Location #116, Villejuif
- Germany (11):
  - Location #90, Augsburg
  - Location #51, Berlin
  - Location #91, Dresden
  - Location #46, Hanover
  - Location #89, Jena
  - Location #50, Kiel
  - Location #111, Ludwigshafen
  - Location #48, Lübeck
  - Location #44, Münster
  - Location #52, Tübingen
  - Location #45, Würzburg
- Israel (3):
  - Location #86, Jerusalem
  - Location #84, Petah Tikva
  - Location #85, Tel Litwinsky
- Italy (5):
  - Location #82, Genoa
  - Location #78, Milan
  - Location #79, Napoli
  - Location #80, Padua
  - Location #81, Siena
- Netherlands (2):
  - Location #59, Groningen
  - Location #60, Leiden
- Poland (2):
  - Location #72, Lubin
  - Location #65, Poznan
- Russia (7):
  - Location #93, Barnaul
  - Location #61, Moscow
  - Location #58, Moscow
  - Location #62, Nizniy Novogrod
  - Location #57, Saint Petersburg
  - Location #94, Samara
  - Location #95, Stavropol
- Spain (3):
  - Location #67, Barcelona
  - Location #54, Valencia
  - Location #68, Zaragoza
- Switzerland (2):
  - Location #118, Bern
  - Location #43, Zurich
- Turkey (Türkiye) (4):
  - Location #122, Ankara
  - Location #124, Antalya
  - Location #121, Izmir
  - Location #123, Kocaeli